CLINICAL TRIAL: NCT05981105
Title: Expanding the Peri-operative Surgical Home Model: ERAS TKR With a Transitional Pain Service (TeleTPS) - Continuous Adductor Canal Catheter Versus Adductor Canal Block for Total Knee Arthroplasty, a Randomized Double-blinded Controlled Trial.
Brief Title: Enhanced Recovery After Major Surgery and Chronic Pain for Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017-1858 pt 2
Record Dates: First submitted 2023-06-16; First posted 2023-08-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Opioid Use; Adductor Canal Block; Total Knee Arthroplasty
MeSH Terms: conditions — Chronic Pain | interventions — Catheters

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized to the intervention group (adductor canal catheter, ACC) or control group (sham adductor canal catheterm, ACB). The research staff and participants will be blinded as to which group the participant is in. The primary investigator and co-investigators will not be blinded. The research staff will provide PI and Co-I with an envelope that informs them which group the participant is randomized to so the proper research activities are carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Adductor Canal Catheter (ACC) - Interventional (Experimental): Patients will received the an adductor canal catheter that continuously infuses numbing medication to their operative leg for 50 hours post-surgery.
  Patients will also communicate with their pain doctor via the Diagnotes application while the catheter is in place.
  Interventions: Device: ambIT pump with catheter
- Adductor Canal Block (ACB) - Control (Sham Comparator): Patients will received the a sham adductor canal catheter that is attached to their operative leg for 50 hours post-surgery.
  Patients will also communicate with their pain doctor via the Diagnotes application while the catheter is in place.
  Interventions: Device: ambIT pump with sham catheter

INTERVENTIONS:
Device: ambIT pump with catheter — 0.2% ropivacaine will be infused through a catheter pump at a rate of 10 ml/hr, 600 ml reservoir.
  Arms: Adductor Canal Catheter (ACC) - Interventional
Device: ambIT pump with sham catheter — sham catheter with no infusion
  Arms: Adductor Canal Block (ACB) - Control

SUMMARY:
The goal of this interventional clinical trial is to assess opioid consumption 24-48 hrs post anesthesia block among patients undergoing total knee arthroplasty. The main question it aims to answer is:

1. Is there a difference in opioid consumption 24-48 hours post block administration among patients that receive an adductor canal catheter (ACC) versus adductor canal block (ACB)?

Participants will be:

* Randomized to receive an adductor canal catheter (ACC) or a sham adductor canal catheter.
* Asked to use the Diagnotes application to communicate with the pain doctor while the catheter is in place.
* Follow up for up to 6 months post-operation. Researchers will compare the interventional group (ACC) to the control group (sham ACC + ACB) to see if there is difference in opioid consumption and chronic pain at 6 months post-operation.

DETAILED DESCRIPTION:
The purpose of this study is to see if adding a continuous ACB catheter will extend analgesia beyond the 24-48 hour period. This interventional clinical trial will assess opioid consumption in patients undergoing total knee arthroplasty 24 to 48 hours after anesthesia block. Rebound pain is a well-known phenomenon in which patients experience severe pain immediately after the nerve block is removed. It is also known that by extending the duration of analgesia, you can reduce or prevent rebound pain. Motor sparing compartment blocks have transformed patients' ability to participate in rehabilitation earlier than ever before, even ambulating on POD 0. Thus, by extending analgesia and encouraging early ambulation, adductor canal catheters are likely to not only reduce opioid consumption but also allow for earlier discharge. The two "hot" themes in recent total knee replacement analgesia pathways are not only providing an effective Enhanced recovery after surgery (ERAD) protocol, but also combating the opioid epidemic through regional anesthesia and non-opioid multimodal pathways. This study will assist in determining which modality is superior (single shot blocks with additive versus catheter) and will introduce a novel method of following patients at home via a transitional pain service (telemedicine). This research will further investigate chronic pain 6 months after surgery.

Patients in the intervention group will have a catheter that continuously infuses numbing medication into their operative leg for 50 hours (up to POD 3). It is hypothesized that the patient will have better pain control, mobility, and less rebound pain, which is common following POD 1. By infusing the catheter with a disposable single use ambIT system (Summit Medical Products), all patients enrolled in the intervention group (ACC) will have the same amount running continuously, allowing the patient to be discharged with the catheter in place before the 50-hour infusion is completed. Prior to discharge, patients will be instructed on how to remove the catheter and will be able to download the Smartphone app "Diagnotes" at the hospital. While the catheter is in place, the Diagnotes app (a HIPPA-compliant text messaging service) will be the patient's primary means of communication with the pain doctor at home.

Patients in the control group will have a sham (fake) catheter attached to their operative leg for 50 hours. Patients will also be instructed on how to remove the catheter prior to discharge and will be able to download the Smartphone app "Diagnotes" in the hospital. While the catheter is in place, the Diagnotes app (a HIPPA-compliant text messaging service) will be the patient's primary means of communication with the pain doctor at home.

Researchers will contact both groups for follow-ups for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for a primary total knee arthroplasty with a participating surgeon
* Age 18 to 75 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (secondary outcomes include questionnaires validated in English only)
* Patients of participating surgeons: Drs. Mayman, Jerabek, Westrich, Su, Della Valle, Alexiades
* Lives within one hour of the hospital
* Has a smartphone

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old and older than 65
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI > 40
* Diabetes
* ASA of III,IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* PCS > 30
* Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)
* Patients with severe valgus deformity or flexion contracture
* Patients unable to follow home catheter instructions and unwilling to go home with an infusing catheter
* Patients who have no home caregivers in the event if a catheter is to be sent home with the patient
* Patients with planned stay at rehab facility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption at 24-48 hours | from 24 hours to 48 hours
  The cumulative opioid consumption 24-48 hours post block administration. Measured in morphine milligram equivalents per day.
  Although collected over a period of time, the total amount will be summed and the average will be reported.

SECONDARY OUTCOMES:
Opioid consumption at 72 hours, 96 hours, and 1 week | 72 hours to 1 week
  The cumulative opioid consumption 72hours, 96 hours, and 1 week post block administration. Measured in morphine milligram equivalents per day.
  Although collected over a period of time, the total amount will be summed and the average will be reported.
Numerical Pain Rating Score | Day of surgery to post operative day (POD) 60
  Patients are asked to give a number between 0 and 10 that best fits their pain intensity. The scale is 0 = 'no pain at all' whereas 10 = 'the worst pain ever possible'.
  Measured at multiple time points: DOS, post-operative day (POD) 1, POD 2, POD 3, POD 4, POD 7, & POD 60
Physical Therapy Milestones | post operative day (POD) 1 up to POD 4
  Collected from the physical therapy notes. This outcome will assess for time to ambulation (measured in distance traveled, stairs, time of ambulating > 30 meters, and reaching discharge criteria).
Patient Satisfaction with Pain Control | post operative day (POD) 1, 2, 4 & 60
  Patients are asked to report on their satisfaction with pain control on a scale of 0 to 10, with 0 = extremely dissatisfied and 10 = extremely satisfied.
Hospital Length of Stay | up to 7 days after the day of surgery
  From when the patient is in the PACU to when the patient has been discharged from the hospital. PACU time = "PACU Transfer In" and Discharge time = "Discharge"
Opioid Related Symptom Distress Scale (ORSDS) | after the surgery end time, on post operative day (POD) 1, 4, and 60
  The Opioid-Related Symptom Distress Scale (ORSDS) is a 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 12 symptoms. The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS is the average of 12 symptom-specific scores.
Number of participants who experienced Buckling/Falls/Quadricep during physical therapy | On post operative day (POD) 1, 2, 3, 4
  Whether a participant experiences buckling, falls, or quadricep weakness during physical therapy, precluding ambulation.
Incidents of participants experiencing a blood loss during surgical procedure | During surgery
  Whether the participant experienced any blood loss during their surgical procedure.
  Measured in binary responses (yes/no).
Block resolution | Up to post operative day 3
  The patient will be asked in the morning of POD 1 when they feel the block has worn off, and in the evening of POD 3 after the catheter has been removed.
Distance of ambulation | post operative day (POD) 0,1,2,3,4
  The total distance of ambulation during physical therapy while the patient is inpatient, collected from the physical therapy notes.
Catheter related complications | up to post operative day 4
  Patient will be asked if they have experience any of the following with regards to the catheter:
  delayed weakness, unintentional dislodgment, leakage, catheter infection, dysesthesias, falls, LAST
Incidences of participants readmitted for pain control | 3 month after surgery
  Whether the patient was readmitted to a hospital for additional pain control.
Block complications | up to post operative day 4
  Patients will report if they experience any block complications including, neuropraxia (saphenous), transient palsies: peroneal, tibial nerve.
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | before surgery and up to post operative day 60
  The survey asks for patients' view about their knee, such as how they feel about their knee and how well they are able to do usual activities. Choices on each question are: none, mild, moderate, severe, extreme
Orthopedic Outcome Flexion/Knee Society Score | 6 weeks
  Patient will be asked about their range of motion (flexion ROM and Extension ROM). Data collected from surgeon's note
SF-36 questionnaire | up to post operative day 60
  The SF-36 measures includes the following: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH).
  Measured on a scale of 1 to 3, with 1 = "yes limited a lot", 2 = "yes limited a little", 3 = "no not limited at all".
  The total score for each participant is calculated and then all the scores are average across all participants.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | at 3 months & 6 months
  The Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (LANSS) comprises of a 7-item pain scale, including the sensory descriptors and items for sensory examination.
  Out of the seven items in the Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (LANSS), five are symptom related and two are examination items.
  If patient reports surgery-related pain greater than 3 on the NRS at the 3 months and 6 months postoperative visit, patient will complete this questionnaire.
Current opioid misuse measure (COMM) | at 3 months & 6 months
  The Current Opioid Misuse Measure (COMM) is a commonly used self-report instrument to identify and monitor aberrant opioid-related behavior in chronic pain patients on opioid therapy.
  At the 3 months and 6 months postoperative visit, if patients are still being prescribed opioids, patient will be asked to fill out the questionnaire
  Choices on the questionnaire are:
  never, seldom, sometimes, often, very often
Incidence of patient contact via text messaging/video calls | up to post operative day 4
  Research staff will mark if patients contacted the pain doctor via the Diagnotes application.
Number of unused opioids | up to post operative day 7
  Patients will be asked at 1 week post-operation, about their pain medication usage (how many pills of your opioid medication do you have left?)
Pain catastrophizing scale (PCS) | before the surgery and up to post operative day 60
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking due to low back pain according to 3 components: rumination, magnification, and helplessness. It is a 13-item scale, with a total range of 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
Pain Disability Index (PDI) | 3 months & 6 months
  The Pain Disability Index (PDI) is a widely-used instrument to measure pain-related disability.
  Scoring: Scores are assigned based on an 11-point scale ranging from 0 (no disability) to 10 (total disability). Scores range from 0 to 70. The higher the index the greater the person's disability due to pain.
Blinding Assessment | up to post operative day 2
  Patient and research staff will report which group they believe the patient was randomized to.
Incidents of participants experiencing block complications | up to post operative day 4
  Data on whether patient experienced quadriceps weakness and foot drop during physical therapy. Collected from physical therapy notes.
Non Opioid Pain medications consumption | up to post operative day 60
  Research staff will document any non-opioid pain medications (lyrica, robaxin, tyelnol, etc) taken by each participant. Medications may be given at the discretion of the APS service.
Intravenous patient control analgesia (IV PCA) usage | up to post operative day 7
  Research staff will document if patient received IV PCA during their stay at the hospital. Measured in morphine equivalent.
  Discharge times can vary from participant to participant (from POD 0 up until POD 2)
Length of induction | During the surgical procedure
  The time it takes for the patient to be induced. Measured from induction start to induction end.
  Times for each participants will be calculated (in minutes) and then average across all participants.
Length of tourniquet use | During the surgical procedure
  The total time to use a tourniquet. Measured from tourniquet inflated time tourniquet deflated time.
  Times for each participants will be calculated (in minutes) and then average across all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Memtsoudis, MD/PhD, Principal Investigator — Hospital for Special Surgery, New York; Jashvant Poeran, MD/PhD, Study Director — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Result] Katz J, Weinrib A, Fashler SR, Katznelzon R, Shah BR, Ladak SS, Jiang J, Li Q, McMillan K, Santa Mina D, Wentlandt K, McRae K, Tamir D, Lyn S, de Perrot M, Rao V, Grant D, Roche-Nagle G, Cleary SP, Hofer SO, Gilbert R, Wijeysundera D, Ritvo P, Janmohamed T, O'Leary G, Clarke H. The Toronto General Hospital Transitional Pain Service: development and implementation of a multidisciplinary program to prevent chronic postsurgical pain. J Pain Res. 2015 Oct 12;8:695-702. doi: 10.2147/JPR.S91924. eCollection 2015. PMID 26508886
- [Result] Chen YK, Boden KA, Schreiber KL. The role of regional anaesthesia and multimodal analgesia in the prevention of chronic postoperative pain: a narrative review. Anaesthesia. 2021 Jan;76 Suppl 1(Suppl 1):8-17. doi: 10.1111/anae.15256. PMID 33426669
- [Result] Benthien JP, Huebner D. Efficacy of continuous catheter analgesia of the sciatic nerve after total knee arthroplasty. Swiss Med Wkly. 2015 Feb 19;145:w14119. doi: 10.4414/smw.2015.14119. eCollection 2015. PMID 25695308
- [Result] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Result] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Result] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Result] Kovalak E, Dogan AT, Uzumcugil O, Obut A, Yildiz AS, Kanay E, Tuzuner T, Ozyuvaci E. A comparison of continuous femoral nerve block and periarticular local infiltration analgesia in the management of early period pain developing after total knee arthroplasty. Acta Orthop Traumatol Turc. 2015;49(3):260-6. doi: 10.3944/AOTT.2015.14.0263. PMID 26200404
- [Result] Horn BJ, Cien A, Reeves NP, Pathak P, Taunt CJ Jr. Femoral Nerve Block vs Periarticular Bupivacaine Liposome Injection After Primary Total Knee Arthroplasty: Effect on Patient Outcomes. J Am Osteopath Assoc. 2015 Dec;115(12):714-9. doi: 10.7556/jaoa.2015.146. PMID 26618816
- [Result] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT05981105/Prot_SAP_000.pdf